CLINICAL TRIAL: NCT01890265
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety and Efficacy of FG-3019 in Patients With Idiopathic Pulmonary Fibrosis
Brief Title: Evaluate the Safety and Efficacy of FG-3019 (Pamrevlumab) in Participants With Idiopathic Pulmonary Fibrosis (IPF)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kyntra Bio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FGCL-3019-067
Record Dates: First submitted 2013-06-24; First posted 2013-07-01 (Estimated); Results first posted 2020-09-04 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-08

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Idiopathic Pulmonary Fibrosis; IPF; Idiopathic Interstitial Pneumonia; Interstitial Lung Disease; Lung Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Idiopathic Interstitial Pneumonias; Lung Diseases, Interstitial; Pulmonary Fibrosis | interventions — pamrevlumab; Immunoglobulin G; nintedanib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, Investigators, and study staff were blinded to treatment assignments and did not have access to the randomization codes. The high-resolution computed tomography (HRCT) readers were blinded to treatment assignments.
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Pamrevlumab (Experimental): Participants will receive pamrevlumab 30 milligram/kilogram (mg/kg) by intravenous (IV) infusion every 3 weeks for a total of 16 infusions over 45 weeks.
  Interventions: Drug: Pamrevlumab
- Placebo (Placebo Comparator): Participants will receive placebo matching pamrevlumab by IV infusion every 3 weeks for a total of 16 infusions over 45 weeks.
  Interventions: Drug: Placebo
- Sub-Study: Pamrevlumab+Pirfenidone or Nintedanib (Active Comparator): Participants will receive pamrevlumab by IV infusion every 3 weeks for a total of 8 infusions over 21 weeks. Initial treatment with pamrevlumab in all active comparator participants will be administered at a dose of 15 mg/kg for the first 2 dose administrations. If these are well tolerated, all following study drug administrations will be at 30 mg/kg.
  Pirfenidone or nintedanib will be dosed according to the instructions in their respective labels and the prescribing physician.
  Interventions: Drug: Pamrevlumab; Drug: Sub-Study: Pirfenidone; Drug: Sub-Study: Nintedanib
- Sub-Study: Placebo+Pirfenidone or Nintedanib (Placebo Comparator): Participants will receive placebo matching pamrevlumab by IV infusion every 3 weeks for a total of 8 infusions over 21 weeks. Initial treatment with placebo in all active comparator participants will be administered at a dose of 15 mg/kg for the first 2 dose administrations. If these are well tolerated, all following study drug administrations will be at 30 mg/kg.
  Pirfenidone or nintedanib will be dosed according to the instructions in their respective labels and the prescribing physician.
  Interventions: Drug: Placebo; Drug: Sub-Study: Pirfenidone; Drug: Sub-Study: Nintedanib

INTERVENTIONS:
Drug: Pamrevlumab — Solution for infusion
  Other Names: Fully human recombinant immunoglobulin G (IgG), kappa monoclonal anti-body.; FG-3019
  Arms: Pamrevlumab; Sub-Study: Pamrevlumab+Pirfenidone or Nintedanib
Drug: Placebo — Solution for infusion
  Arms: Placebo; Sub-Study: Placebo+Pirfenidone or Nintedanib
Drug: Sub-Study: Pirfenidone — Pirfenidone concomitant therapy will not be provided by the Sponsor.
  Other Names: Esbeiet
  Arms: Sub-Study: Pamrevlumab+Pirfenidone or Nintedanib; Sub-Study: Placebo+Pirfenidone or Nintedanib
Drug: Sub-Study: Nintedanib — Nintedanib concomitant therapy will not be provided by the Sponsor.
  Other Names: Ofev
  Arms: Sub-Study: Pamrevlumab+Pirfenidone or Nintedanib; Sub-Study: Placebo+Pirfenidone or Nintedanib

SUMMARY:
To evaluate the safety and tolerability of pamrevlumab in participants with IPF, and the efficacy of pamrevlumab in slowing the loss of forced vital capacity (FVC) and the progression of IPF in these participants.

DETAILED DESCRIPTION:
The study has been amended in February 2016 to further allow for the enrollment of a subgroup of participants (N=60) who will be allowed to receive treatment with approved IPF therapy with pirfenidone or with nintedanib as concomitant therapy.

These additional participants will be stratified by background therapy, randomized to pamrevlumab or placebo, and followed up for 24 weeks. The main objective of the study remains safety. Pharmacokinetic (PK) samples to assess drug concentrations will also be collected.

This sub-study portion only applies to a select United States centers.

Enrollment for the main study was completed on 29 June 2016. Enrollment for the sub-study was completed on 16 December 2016.

ELIGIBILITY:
Inclusion Criteria:

1. Age 40 to 80 years, inclusive.
2. Diagnosis of IPF as defined by current international guidelines. Each participant must have 1 of the following: (1) Usual Interstitial Pneumonia (UIP) Pattern on an available high-resolution computed tomography (HRCT) scan; or (2) Possible UIP Pattern on an available HRCT scan and surgical lung biopsy within 4 years of Screening showing UIP Pattern.
3. History of IPF of ≤5 years duration with onset defined as the date of the first diagnosis of IPF by HRCT or surgical lung biopsy.
4. Interstitial pulmonary fibrosis defined by HRCT scan at Screening, with evidence of ≥10% to <50% parenchymal fibrosis (reticulation) and <25% honeycombing, within the whole lung, as determined by the HRCT central reader.
5. FVC percent of predicted value ≥55% at Screening.
6. Female participants of childbearing potential (including those <1 year postmenopausal) must be willing to use a medically acceptable method of contraception, for example, an oral contraceptive, depot progesterone, or intrauterine device. Male participants with female partners of childbearing potential who are not using birth control as described above must use a barrier method of contraception (for example, condom) if not surgically sterile (for example, vasectomy).
7. For sub-study only: Receiving treatment for IPF with a stable dose of pirfenidone or with a stable dose of nintedanib for at least 3 months before Screening initiation and willing to continue treatment with pirfenidone or with nintedanib according to the corresponding approved label and the prescribing physician, including all listed safety requirements (for example, liver function tests, avoidance of sunlight and sunlamp exposure and wearing of sunscreen and protective clothing daily for pirfenidone, and smoking cessation).

Exclusion Criteria:

1. Women who are pregnant or nursing.
2. Infiltrative lung disease other than IPF, including any of the other types of idiopathic interstitial pneumonias (Travis, 2013); lung diseases related to exposure to fibrogenic agents or other environmental toxins or drugs; other types of occupational lung diseases; granulomatous lung diseases; pulmonary vascular diseases; systemic diseases, including vasculitis and connective tissue diseases.
3. HRCT scan findings at Screening are inconsistent with UIP Pattern, as determined by the HRCT central reader.
4. Pathology diagnosis on surgical lung biopsy is anything other than UIP Pattern, as determined by the local pathologist.
5. The Investigator judges that there has been sustained improvement in the severity of IPF during the 12 months prior to Screening, based on changes in FVC, diffusing capacity of the lung for carbon monoxide (DLCO), and/or HRCT scans of the chest.
6. Clinically important abnormal laboratory tests.
7. Upper or lower respiratory tract infection of any type within 4 weeks of the first Screening visit.
8. Acute exacerbation of IPF within 3 months of the first Screening visit.
9. Use of medications to treat IPF within 5 half-lives of Day 1 dosing. If monoclonal antibodies were used, the last dose of the antibody must be at least 4 weeks before Day 1 dosing. This applies to participants enrolled in Main Study only.
10. Use of any investigational drugs, including any investigational drugs for IPF, within 4 weeks prior to Day 1 dosing.
11. History of cancer diagnosis of any type in the 3 years preceding Screening, excluding non-melanomatous skin cancer, localized bladder cancer, or in situ cancers.
12. Diffusing capacity (DLCO) less than 30% of predicted value.
13. History of allergic or anaphylactic reaction to human, humanized, chimeric, or murine monoclonal antibodies.
14. Previous treatment with FG-3019.
15. Body weight greater than 130 kilograms.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2013-07-30 (Actual); Primary Completion 2017-11-16 (Actual); Study Completion 2017-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Wencel, M.D, Principal Investigator — Via Christi Clinic, P.A., USA; Joao de Andrade, M.D, Principal Investigator — The Kirklin Clinic, USA; Peter LaCamera, M.D., Principal Investigator — Steward St. Elizabeth's Medical Center, USA; Danielle Antin-Ozerkis, M.D., Principal Investigator — Yale University, USA; Rishi Raj, M.D., Principal Investigator — Northwestern University; Neil Ettinger, M.D, Principal Investigator — St Luke's Hospital, USA; Rafael Perez, M.D, Principal Investigator — University of Louisville, USA; Timothy Albertson, M.D, Principal Investigator — University of California Davis Medical Center, USA; Yolanda Mageto, M.D., Principal Investigator — Vermont Lung Center, USA; Srihari Veeraraghavan, M.D, Principal Investigator — Emory University, USA; Nishant Gupta, M.D, Principal Investigator — University of Cinncinati, USA; Kevin Gibson, M.D, Principal Investigator — University of Pittsburgh Medical Center, USA; Lisa Lancaster, M.D., Principal Investigator — Vanderbilt University, USA; Mary Beth Scholand, M.D., Principal Investigator — University of Utah - Lung Health Research, USA; Mark Hamblin, M.D., Principal Investigator — University of Kansas Medical Center, USA; John Fitzgerald, M.D., Principal Investigator — University of Texas Southwestern Medical Center, USA; John Belperio, M.D., Principal Investigator — David Geffen School of Medicine at UCLA, USA; Richard Enelow, M.D., Principal Investigator — Dartmouth-Hitchcock Medical Center, USA; Evans R Fernandez-Perez, M.D, Principal Investigator — National Jewish Center, USA; Peter A Bercz, M.D, Principal Investigator — Pensacola Research Consultants, INC., USA; Krishna Thavarajah, M.D., Principal Investigator — Henry Ford Medical Center, USA; James Britt, M.D., Principal Investigator — University of Maryland, College Park; Danielle D. Hosmer, Principal Investigator — Legacy Research Institute, USA; David Lederer, M.D., Principal Investigator — Columbia University Medical Center, USA; Murali Ramaswamy, M.D., Principal Investigator — PulmonIx LLC, USA; Thomas O'Brien, M.D., Principal Investigator — Pulmonary Disease Specialist, PA, USA; Nadim Srour, M.D., Principal Investigator — Université de Sherbrooke / Hôpital Charles LeMoyne, Canada; Elvis Irusen, M.D., Principal Investigator — Tygerberg Hospital Respiratory Research Unit, South Africa; Anish Ambaram, M.D., Principal Investigator — Life Mount Edgecombe Hospital, South Africa; Heidi Siebert, M.D., Principal Investigator — Into Research, South Africa; Elizabeth Veitch, M.D., Principal Investigator — Concord Repatriation, Australia; Huw Davies, M.D., Principal Investigator — Daw Park Repatriation, Australia; Lutz Beckert, M.D., Principal Investigator — Christchurch Hospital NZ, New Zealand; Catherina Chang, M.D., Principal Investigator — Waikato Hospital, New Zealand; Benedict Brockway, M.D., Principal Investigator — Dunedin Public Hospital, New Zealand; Suzanne Poole, M.D., Principal Investigator — Tauranga Hospital, New Zealand; Raja Dhar, M.D., Principal Investigator — Fortis Hospitals, India; Bhanu Singh, M.D., Principal Investigator — Midland Healthcare & Research Center, India; Nandagopal Velayuthaswamy, M.D., Principal Investigator — Sri Bala Medical Centre and Hospital, India; Sujeet Rajan, M.D., Principal Investigator — Bhatia Hospital, India; Priya Ramachandran, M.D., Principal Investigator — St Johns Medical College Hospital, India; Natalia Stoeva, M.D., Principal Investigator — MHAT 'Tokuda Hospital Sofia', AD, Department of Pulmonology, Bulgaria
Locations (42):
- United States (26):
  - The Kirklin Clinic, Birmingham, Alabama
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - UC Davis Medical Center, Sacramento, California
  - National Jewish Health, Denver, Colorado
  - Yale University, New Haven, Connecticut
  - Pulmonary Disease Specialist, PA, Kissimmee, Florida
  - Pensacola Research Consultants, Inc., d.b.a. Avanza Medical Research Center, Pensacola, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Via Christi Clinic, P.A., Wichita, Kansas
  - University of Louisville, Louisville, Kentucky
  - University of Maryland, Baltimore, Maryland
  - Steward St. Elizabeth's Medical Center, Boston, Massachusetts
  - Henry Ford Medical Center, Detroit, Michigan
  - St. Luke's Hospital, Chesterfield, Missouri
  - Columbia University Medical Center, New York, New York
  - PulmonIx LLC, Greensboro, North Carolina
  - University of Cinncinati, Cincinnati, Ohio
  - Dartmouth-Hitchcock Medical Center, Lebanon, Ohio
  - Legacy Research Institute, Portland, Oregon
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Utah - Lung Health Research, Salt Lake City, Utah
  - Vermont Lung Center, Colchester, Vermont
- Australia (2):
  - Concord Repatriation, Concord, New South Wales
  - Daw Park Repatriation, Adelaide, South Australia
- MHAT 'Tokuda Hospital Sofia', AD, Department of Pulmonology, Sofia, Bulgaria
- Université de Sherbrooke / Hôpital Charles LeMoyne, Greenfield Park, Quebec, Canada
- India (5):
  - St Johns Medical College Hospital, Bangalore, Karnataka
  - Bhatia Hospital, Mumbai, Maharashtra
  - Sri Bala Medical Centre and Hospital, Coimbatore, Tamil Nadu
  - Midland Healthcare & Research Center, Lucknow, Uttar Pradesh
  - Fortis Hospitals, Kolkata, West Bengal
- New Zealand (4):
  - Christchurch Hospital NZ, Christchurch
  - Dunedin Public Hospital, Dunedin
  - Waikato Hospital, Hamilton
  - Tauranga Hospital, Tauranga
- South Africa (3):
  - Into Research, Pretoria, Gauteng
  - Life Mount Edgecombe Hospital, Durban, KwaZulu-Natal
  - Tygerberg Hospital Respiratory Research Unit, Cape Town, Western Cape

REFERENCES:
- [Background] Lipson KE, Wong C, Teng Y, Spong S. CTGF is a central mediator of tissue remodeling and fibrosis and its inhibition can reverse the process of fibrosis. Fibrogenesis Tissue Repair. 2012 Jun 6;5(Suppl 1):S24. doi: 10.1186/1755-1536-5-S1-S24. eCollection 2012. PMID 23259531
- [Derived] Kim GH, Zhang X, Brown MS, Poole L, Goldin J. Minimum clinically important difference in Quantitative Lung Fibrosis score associated with all-cause mortality in idiopathic pulmonary fibrosis: subanalysis from two phase II trials of pamrevlumab. BMJ Open. 2025 May 12;15(5):e094559. doi: 10.1136/bmjopen-2024-094559. PMID 40355288
- [Derived] Richeldi L, Fernandez Perez ER, Costabel U, Albera C, Lederer DJ, Flaherty KR, Ettinger N, Perez R, Scholand MB, Goldin J, Peony Yu KH, Neff T, Porter S, Zhong M, Gorina E, Kouchakji E, Raghu G. Pamrevlumab, an anti-connective tissue growth factor therapy, for idiopathic pulmonary fibrosis (PRAISE): a phase 2, randomised, double-blind, placebo-controlled trial. Lancet Respir Med. 2020 Jan;8(1):25-33. doi: 10.1016/S2213-2600(19)30262-0. Epub 2019 Sep 28. PMID 31575509

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult participants with a history of idiopathic pulmonary fibrosis (IPF) ≤5 years duration and a forced vital capacity (FVC) predicted value ≥55% at screening were randomized to receive pamrevlumab or placebo.
Pre-assignment Details: This Phase 2 study was conducted at 44 study centers in 7 countries from July 2013 to November 2017.
Groups:
- Pamrevlumab: Participants received pamrevlumab 30 milligram/kilogram (mg/kg) by intravenous (IV) infusion every 3 weeks for a total of 16 infusions over 45 weeks.
- Placebo: Participants received placebo matching pamrevlumab by IV infusion every 3 weeks for a total of 16 infusions over 45 weeks.
- Sub-Study: Pamrevlumab+Pirfenidone: Participants received pamrevlumab by IV infusion every 3 weeks for a total of 8 infusions over 21 weeks. Initial treatment with pamrevlumab in all active comparator participants was administered at a dose of 15 mg/kg for the first 2 dose administrations. If these were well tolerated, all following study drug administrations were at 30 mg/kg.
  Pirfenidone was dosed according to the instructions in the label and the prescribing physician.
- Sub-Study: Placebo+Pirfenidone: Participants received placebo matching pamrevlumab by IV infusion every 3 weeks for a total of 8 infusions over 21 weeks. Initial treatment with placebo in all active comparator participants were administered at a dose of 15 mg/kg for the first 2 dose administrations. If these were well tolerated, all following study drug administrations were at 30 mg/kg.
  Pirfenidone was dosed according to the instructions in the label and the prescribing physician.
- Sub-Study: Pamrevlumab+Nintedanib: Participants received pamrevlumab by IV infusion every 3 weeks for a total of 8 infusions over 21 weeks. Initial treatment with pamrevlumab in all active comparator participants was administered at a dose of 15 mg/kg for the first 2 dose administrations. If these were well tolerated, all following study drug administrations were at 30 mg/kg.
  Nintedanib was dosed according to the instructions in the label and the prescribing physician.
- Sub-Study: Placebo+Nintedanib: Participants received placebo matching pamrevlumab by IV infusion every 3 weeks for a total of 8 infusions over 21 weeks. Initial treatment with placebo in all active comparator participants were administered at a dose of 15 mg/kg for the first 2 dose administrations. If these were well tolerated, all following study drug administrations were at 30 mg/kg.
  Nintedanib was dosed according to the instructions in the label and the prescribing physician.
Period: Overall Study
Arm/Group | Pamrevlumab | Placebo | Sub-Study: Pamrevlumab+Pirfenidone | Sub-Study: Placebo+Pirfenidone | Sub-Study: Pamrevlumab+Nintedanib | Sub-Study: Placebo+Nintedanib
Started | 50 | 53 | 24 | 12 | 15 | 6
Safety Population (Population included randomized participants who received any amount of study medication.) | 50 | 53 | 24 | 12 | 15 | 6
Intent-to-Treat (ITT) Population (Population included participants who were randomized and met all protocol eligibility criteria.) | 50 | 51 | 24 | 12 | 15 | 6
Completed | 40 | 40 | 20 | 12 | 13 | 6
Not Completed | 10 | 13 | 4 | 0 | 2 | 0
Not completed — Other (Unspecified reason) | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Progressive disease | 6 | 6 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 1 | 0 | 0 | 0 | 0
Not completed — Death | 2 | 3 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 3 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Randomized participants who received any amount of study medication (Safety Population).
Groups:
- Pamrevlumab: Participants received pamrevlumab 30 mg/kg by IV infusion every 3 weeks for a total of 16 infusions over 45 weeks.
- Sub-Study:Placebo+Pirfenidone: Participants received placebo matching pamrevlumab by IV infusion every 3 weeks for a total of 8 infusions over 21 weeks. Initial treatment with placebo in all active comparator participants were administered at a dose of 15 mg/kg for the first 2 dose administrations. If these were well tolerated, all following study drug administrations were at 30 mg/kg.
  Pirfenidone was dosed according to the instructions in the label and the prescribing physician.
- Sub-Study:Pamrevlumab+Nintedanib: Participants received pamrevlumab by IV infusion every 3 weeks for a total of 8 infusions over 21 weeks. Initial treatment with pamrevlumab in all active comparator participants was administered at a dose of 15 mg/kg for the first 2 dose administrations. If these were well tolerated, all following study drug administrations were at 30 mg/kg.
  Nintedanib was dosed according to the instructions in the label and the prescribing physician.
- Total: Total of all reporting groups
Arm/Group | Pamrevlumab | Placebo | Sub-Study: Pamrevlumab+Pirfenidone | Sub-Study:Placebo+Pirfenidone | Sub-Study:Pamrevlumab+Nintedanib | Sub-Study: Placebo+Nintedanib | Total
Number analyzed (Participants) | 50 | 53 | 24 | 12 | 15 | 6 | 160
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.3 (7.05) | 68.4 (7.20) | 68.6 (6.27) | 68.4 (5.50) | 71.1 (7.32) | 65.2 (4.62) | 68.5 (6.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 10 | 7 | 4 | 2 | 3 | 43
  Male | 33 | 43 | 17 | 8 | 13 | 3 | 117
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 49 | 52 | 0 | 0 | 0 | 0 | 101
  Not Hispanic or Latino | 1 | 1 | 24 | 12 | 15 | 6 | 59
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 5 | 3 | 0 | 0 | 0 | 0 | 8
  Black or African American | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 41 | 44 | 24 | 12 | 15 | 6 | 142
  Other | 4 | 5 | 0 | 0 | 0 | 0 | 9

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in FVC (Percent of Predicted FVC Value [% Predicted]) to Week 48
Description: FVC in liters was measured during the spirometry assessments at screening and during the randomized treatment period at Day 1 and every 12 weeks. The FVC (% predicted) was calculated for the corresponding gender-race-age group. The least squares (LS) mean change from Baseline to Week 48 (end of the randomized treatment period) in FVC (% predicted) is presented. Baseline was defined as the mean of the last screening visit and the Day 1 visit values. Other statistical analysis data is reported in the statistical analysis section. Observed data from all visits were included in the model.
Time Frame: Baseline (Screening and Day 1), Week 48
Population: Randomized participants who met all protocol eligibility criteria (ITT population). Data for the participants who were included in the pamrevlumab and placebo arms in the Main Study were collected for this Outcome Measure.
Measure: Mean (Standard Error); unit: % predicted FVC
Arm/Group | Pamrevlumab | Placebo
Number analyzed (Participants) | 50 | 51
% predicted FVC
  Baseline | 74.51 (1.682) | 72.82 (1.512)
  Change from Baseline at Week 48 | -2.71 (0.624) | -7.20 (1.664)
Statistical Analysis 1: Comparison: Pamrevlumab vs Placebo; The absolute LS mean treatment difference (pamrevlumab - placebo) for change from Baseline to Week 48 in FVC (% predicted) is presented; Test type: Superiority; p = 0.0331, Random coefficient regression — The analysis of the change from Baseline to Week 48 in FVC (% predicted) was based on the random coefficient regression model based on observed cases; LS mean difference = 4.33, 95% CI 2-sided [0.35 to 8.3]

2. Secondary Outcome: Mean Change From Baseline in the HRCT Quantitative Lung Fibrosis (QLF) Score to Week 24 and Week 48
Description: The extent of pulmonary fibrosis was measured by HRCT scans of the chest at screening and at Weeks 24 and 48, to determine the HRCT QLF score. Each lung was divided into 5 lobes (right upper, right middle, right lower, left upper, left lower). For the quantitative HRCT analyses, a computer read the images and quantified the percent (%) and volume (mL) of fibrosis for the whole lung by averaging the scores from each of 5 lung lobes. Baseline was defined as the Screening evaluation. Missing data were imputed using the multiple imputation (MI) method to handle missing values.
Time Frame: Baseline (Screening), Week 24 and Week 48
Population: Randomized participants who met all protocol eligibility criteria (ITT population) and who also had a baseline fibrosis evaluation. Data for the participants who were included in the pamrevlumab and placebo arms in the Main Study were collected for this Outcome Measure.
Measure: Mean (Standard Error); unit: Percent of fibrosis
Arm/Group | Pamrevlumab | Placebo
Number analyzed (Participants) | 47 | 49
Percent of fibrosis
  Baseline | 13.9 (1.44) | 14.7 (1.09)
  Change from Baseline at Week 24 | 0.8 (0.34) | 2.6 (0.55)
  Change from Baseline at Week 48 | 2.7 (0.47) | 6.0 (1.15)
Statistical Analysis 1: Comparison: Pamrevlumab vs Placebo; The absolute LS mean treatment difference (pamrevlumab - placebo) for change from Baseline to Week 24 in QLF score is presented; Test type: Superiority; p = 0.0236, ANCOVA with MI; LS mean difference = -1.8, 95% CI 2-sided [-3.3 to -0.2]
Statistical Analysis 2: Comparison: Pamrevlumab vs Placebo; The absolute LS mean treatment difference (pamrevlumab - placebo) for change from Baseline to Week 48 in QLF score is presented; Test type: Superiority; p = 0.0729, ANCOVA with MI; LS mean difference = -3.2, 95% CI 2-sided [-6.6 to 0.3]

3. Secondary Outcome: Number of Participants With IPF Progression Events up to Week 48
Description: IPF progression events included death from any cause or absolute decline in FVC (% predicted) value of ≥10%, confirmed by repeat spirometry. Classification of FVC (% predicted) declined ≥10% was based on observed and imputed data. Missing data in FVC (% predicted) were imputed using the predicted values from the random coefficient module with treatment, visit, visit-by-treatment interaction, and Baseline FVC (% predicted) as fixed effects and linear slope as random effect.
Time Frame: Baseline (Screening and Day 1) up to Week 48
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Pamrevlumab | Placebo
Number analyzed (Participants) | 50 | 51
Participants | 5 | 16
Statistical Analysis 1: Comparison: Pamrevlumab vs Placebo; The absolute treatment difference (pamrevlumab - placebo) for percentage of participants with IPF progression at Week 48 is presented; Test type: Superiority; p = 0.0133, Regression, Logistic; Absolute difference = -21.4, 95% CI 2-sided [-36.6 to -6.2]

4. Secondary Outcome: Mean Change From Baseline in the Health-Related Quality of Life (HRQoL) Saint George's Respiratory Questionnaire (SGRQ) Domain and Total Scores to Week 24 and Week 48
Description: HRQoL was assessed by the SGRQ to measure health impairment, and includes 17 questions in 3 domains: Symptoms, Activity and Impacts. The domain and total scores range from 0 to 100, with 0 indicating the best and 100 indicating the worst possible health status. Missing data at post-baseline visits were imputed as the predicted values from the random coefficient model which included treatment, visit, visit-by-treatment interaction, and Baseline SGRQ score as fixed effects and linear slope of visit as random effect.
Time Frame: Baseline (Day 1), Week 24 and Week 48
Population: Randomized participants who met all protocol eligibility criteria (ITT population) and who also had a baseline and at least 1 follow-up value. Data for the participants who were included in the pamrevlumab and placebo arms in the Main Study were collected for this Outcome Measure.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Pamrevlumab | Placebo
Number analyzed (Participants) | 47 | 46
score on a scale
  Symptoms Score at Baseline | 48.32 (3.194) | 50.43 (2.579)
  Symptoms Score Change from Baseline at Week 24 | -0.36 (2.045) | -1.74 (2.205)
  Symptoms Score Change from Baseline at Week 48 | -3.06 (2.336) | 1.56 (2.675)
  Activity Score at Baseline | 55.69 (4.038) | 60.46 (2.803)
  Activity Score Change from Baseline at Week 24 | -0.05 (1.889) | 0.26 (1.948)
  Activity Score Change from Baseline at Week 48 | -4.06 (2.432) | 1.35 (2.599)
  Impacts Score at Baseline | 31.38 (3.361) | 31.28 (2.766)
  Impacts Score Change from Baseline at Week 24 | -1.08 (1.518) | -0.50 (2.238)
  Impacts Score Change from Baseline at Week 48 | -1.77 (2.306) | 3.04 (3.106)
  Total Score at Baseline | 41.75 (3.229) | 43.55 (2.390)
  Total Score Change from Baseline at Week 24 | -0.63 (1.220) | -0.73 (1.899)
  Total Score Change from Baseline at Week 48 | -2.75 (1.729) | 2.46 (2.719)

5. Secondary Outcome: Number of Participants With a Respiratory-Related Hospitalization
Description: Respiratory-related hospitalizations were reported by participants and recorded by the Investigators.
Time Frame: Week 55
Population: Randomized participants who received any amount of study medication (Safety Population). Data for the participants who were included in the pamrevlumab and placebo arms in the Main Study were collected for this Outcome Measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Pamrevlumab | Placebo
Number analyzed (Participants) | 50 | 53
Participants | 5 | 7

6. Secondary Outcome: Number of Participants With a Respiratory-Related Death
Description: Investigators determined whether a death was respiratory-related.
Time Frame: Week 55
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Pamrevlumab | Placebo
Number analyzed (Participants) | 50 | 53
Participants | 2 | 3

7. Secondary Outcome: Number of Participants With No Decline in FVC (% Predicted) at Week 48
Description: FVC in liters was measured during the spirometry assessments. The FVC (% predicted) was calculated for the corresponding gender-race-age group. Baseline was defined as the mean of the last screening visit and the Day 1 visit values. Classification of 'No decline' is based on observed and imputed data. Missing data in FVC (% predicted) are imputed using the predicted values from the random coefficient model with treatment, visit, visit-by-treatment interaction, and Baseline FVC (% predicted) as fixed effects and linear slope of visit as random effect.
Time Frame: Baseline (Day 1) to Week 48.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Pamrevlumab | Placebo
Number analyzed (Participants) | 50 | 51
Participants | 11 | 13

ADVERSE EVENTS:
Time Frame: Day 1 up to Week 49
Description: Randomized participants who received any amount of study medication (Safety Population).
Arm/Group | Pamrevlumab | Placebo | Sub-Study: Pamrevlumab+Pirfenidone | Sub-Study: Placebo+Pirfenidone | Sub-Study: Pamrevlumab+Nintedanib | Sub-Study: Placebo+Nintedanib
All-Cause Mortality (participants affected / at risk) | 2/50 | 3/53 | 1/24 | 0/12 | 0/15 | 0/6
Serious Adverse Events (participants affected / at risk) | 12/50 | 8/53 | 2/24 | 1/12 | 0/15 | 1/6
Other Adverse Events (participants affected / at risk) | 42/50 | 41/53 | 19/24 | 12/12 | 14/15 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pamrevlumab (N=50) | Placebo (N=53) | Sub-Study: Pamrevlumab+Pirfenidone (N=24) | Sub-Study: Placebo+Pirfenidone (N=12) | Sub-Study: Pamrevlumab+Nintedanib (N=15) | Sub-Study: Placebo+Nintedanib (N=6)
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 (0) | 2 (2) | 0 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0
Mesenteric haematoma (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0
Antisynthetase syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (5) | 1 | 0 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 | 0 | 0 | 0
Peripheral artery aneurysm (Vascular disorders) | 0 (0) | 1 (1) | 0 | 0 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0) | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pamrevlumab (N=50) | Placebo (N=53) | Sub-Study: Pamrevlumab+Pirfenidone (N=24) | Sub-Study: Placebo+Pirfenidone (N=12) | Sub-Study: Pamrevlumab+Nintedanib (N=15) | Sub-Study: Placebo+Nintedanib (N=6)
Aortic valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Aortic valve sclerosis (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cardiac aneurysm (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Left atrial dilatation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Right atrial dilatation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 3 | 0 | 0 | 0 | 0
Tricuspid valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 4 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 4 | 1 | 1 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 8 | 4 | 1 | 2 | 3 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Gingival swelling (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 7 | 7 | 0 | 1 | 0 | 2
Retching (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Effusion (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Feeling cold (General disorders) | 0 | 0 | 0 | 1 | 1 | 0
Feeling hot (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Chest discomfort (General disorders) | 3 | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 4 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 10 | 4 | 3 | 1 | 1 | 0
Oedema peripheral (General disorders) | 4 | 2 | 0 | 0 | 1 | 0
Pain (General disorders) | 4 | 0 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 2 | 6 | 2 | 1 | 3 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0
Respiratory tract infection (Infections and infestations) | 15 | 10 | 2 | 3 | 1 | 1
Sinusitis (Infections and infestations) | 8 | 8 | 0 | 0 | 0 | 3
Urinary tract infection (Infections and infestations) | 10 | 4 | 1 | 1 | 1 | 1
Viral infection (Infections and infestations) | 0 | 5 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 3 | 1 | 0 | 0 | 0
Face injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Scratch (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Blood iron decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Blood potassium increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Electrophoresis protein abnormal (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Heart sounds abnormal (Investigations) | 3 | 0 | 0 | 0 | 0 | 0
Oxygen consumption increased (Investigations) | 0 | 3 | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 2 | 0 | 0 | 1 | 1
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 5 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 2 | 1 | 1 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Basosquamous carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 4 | 0 | 1 | 2 | 1 | 0
Headache (Nervous system disorders) | 4 | 6 | 1 | 2 | 0 | 0
Hypogeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Migraine (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Sacral radiculopathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 3 | 5 | 1 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 4 | 1 | 1 | 1 | 0 | 0
Calculus bladder (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Crystalluria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 3 | 0 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 14 | 23 | 3 | 3 | 2 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 | 11 | 2 | 2 | 3 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 10 | 7 | 4 | 0 | 2 | 0
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 9 | 5 | 5 | 3 | 4 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 1 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 0 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0 | 2 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 0 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 0 | 0 | 0 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Precancerous skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Tooth extraction (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0 | 0
Flushing (Vascular disorders) | 3 | 4 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 3 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (3):
  • Study Protocol (2016-12-12): https://cdn.clinicaltrials.gov/large-docs/65/NCT01890265/Prot_000.pdf
  • Statistical Analysis Plan: Part 1 (2017-07-26): https://cdn.clinicaltrials.gov/large-docs/65/NCT01890265/SAP_001.pdf
  • Statistical Analysis Plan: Part 2 (2018-03-14): https://cdn.clinicaltrials.gov/large-docs/65/NCT01890265/SAP_002.pdf